CLINICAL TRIAL: NCT01135589
Title: Efficacy and Safety in Micafungin Sodium for Prophylaxis Against Invasive Fungal Disease During Neutropenia in Pediatric & Adolescent Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Micafungin Prevention Study for Fungal Disease in Child Receiving Allogenic Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Director, Astellas Pharma, Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KSPHO 2010-02
Record Dates: First submitted 2010-05-25; First posted 2010-06-03 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-06

CONDITIONS: Neutropenia; Hematopoietic Stem Cell Transplantation; Invasive Fungal Disease
Keywords: pediatric; adolescent; micafungin
MeSH Terms: conditions — Neutropenia; Invasive Fungal Infections | interventions — Micafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HSCT (Experimental)
  Interventions: Drug: Micafungin

INTERVENTIONS:
Drug: Micafungin — i.v.
  Other Names: FK463; Fungard

SUMMARY:
This study is to evaluate safety and prophylaxis effect of micafungin after hematopoietic stem cell transplantation. Micafungin is administered until confirmation of neutrophil engraftment or treatment failure.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate absence of proven, probable, possible, suspected invasive fungal disease (IFDs) through the end of prophylaxis therapy and during 4 weeks after stopping of micafungin prophylaxis after allogeneic hematopoietic stem cell transplantation in pediatric and adolescent neutropenia patients. Patients will receive micafungin until the earliest of the following: 1) neutrophil engraftment; 2) development of proven, provable, possible or suspected invasive fungal disease; 3) development of unacceptable drug toxicity; 4) withdrawal from study participation or discontinuation of study treatment. Safety profile of micafungin is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients will receive allogeneic hematopoietic stem cell transplantation

Exclusion Criteria:

* Aspartate transaminase or alanine transaminase level > 5 times UNL
* Bilirubin > 2. 5 times UNL
* History of allergy, sensitivity, or any serious reaction to an echinocandin
* Invasive fungal disease at the time of enrolment
* Systemic antifungal therapy within 72 hrs before administration of the first dose of study drug
* Positive pregnancy test

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 145 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Absence rate of IFDs assessed by physical examination and serum galactomannan test | during micafungin prophylaxis therapy and during 4 weeks after stopping of micafungin prophylaxis

SECONDARY OUTCOMES:
Survival rate | at day 100
Safety assessed by lab-test and adverse events | during micafungin prophylaxis therapy

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (7):
- South Korea (7):
  - Busan
  - Daegu
  - Daejeon
  - Goyang
  - Hwasun
  - Seoul
  - Suwon